CLINICAL TRIAL: NCT00000961
Title: A Phase II Study to Evaluate the Safety, Tolerance and Efficacy of Hyperimmune Anti-HIV Intravenous Immunoglobulin (HIVIG) and of Zidovudine (ZDV) in Infants With Documented HIV Infections
Brief Title: The Safety and Effectiveness of Hyperimmune Anti-HIV Intravenous Immunoglobulin (HVIG) Plus Zidovudine in HIV-Infected Infants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Abbott (Industry); Glaxo Wellcome (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 131
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine

INTERVENTIONS:
Drug: Anti-HIV Immune Serum Globulin (Human)
Drug: Zidovudine

SUMMARY:
To determine the safety and tolerance of hyperimmune anti-HIV intravenous immunoglobulin (HIVIG) and of zidovudine (AZT) in infants with established HIV infection; to get preliminary evidence for the effectiveness of this type of treatment in preventing the advance of disease in HIV infected infants. HIVIG may be an effective agent that either alone or in combination with AZT will prevent progression of clinical disease.

DETAILED DESCRIPTION:
HIVIG may be an effective agent that either alone or in combination with AZT will prevent progression of clinical disease.

Participants are randomized to receive either oral AZT or HIVIG. Patients may receive treatment for a maximum of 48 weeks. Patients are evaluated during treatment at weeks 2, 4, and every 4 weeks thereafter. Infants who are receiving HIVIG initially are treated with the appropriate age-adjusted dose of oral AZT in addition to HIVIG if they meet clinical disease progression criteria. All participants who have completed 48 weeks of treatment or who are discontinued from treatment are followed every 3 months for an additional 48 weeks. This follow-up may be conducted over the telephone.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Recommended:
* Standard immunizations. Should repeat MMR 3 months after discontinuing study.
* Benadryl and/or aspirin.
* Pneumocystis carinii pneumonia prophylaxis.
* Systemic ketoconazole and acyclovir, or oral nystatin for acute therapy.
* Aerosol ribavirin for short-term treatment of RSV.

Concurrent Treatment:

Allowed:

* Blood transfusion.

Patients must have the following:

* Parent or guardian available to give written informed consent.
* Protocol requires prior Institutional Review Board (IRB) approval before any subject is entered into study.

Prior Medication:

Allowed:

* Gammaglobulin, intravenous (IV) or intramuscular (IM).
* Immunoglobulin, IV (IVIG).
* Maternal antiretroviral treatment during pregnancy.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Symptomatic of any class P-2 symptoms (except lymphadenopathy at time of study entry.
* Presence of serious acute infection requiring parenteral treatment at time of study entry.

Concurrent Medication:

Excluded:

* Prophylaxis for oral candidiasis or otitis media or other infections.
* Immunoglobulin therapy (except single dose or for hypogammaglobulinemia).
* Ketoconazole, acyclovir, or nystatin for prophylaxis.

Patients with the following are excluded:

* Symptomatic of any class P-2 symptoms (except lymphadenopathy at time of study entry.
* Presence of serious acute infection requiring parenteral treatment at time of study entry.

Prior Medication:

Excluded:

* Antiretroviral treatment or experimental treatment within 2 weeks of entry.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112
Dates: Primary Completion 1991-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connor E, Study Chair

REFERENCES:
- [Background] Spector SA, Gelber RD, McGrath N, Wara D, Barzilai A, Abrams E, Bryson YJ, Dankner WM, Livingston RA, Connor EM. A controlled trial of intravenous immune globulin for the prevention of serious bacterial infections in children receiving zidovudine for advanced human immunodeficiency virus infection. Pediatric AIDS Clinical Trials Group. N Engl J Med. 1994 Nov 3;331(18):1181-7. doi: 10.1056/NEJM199411033311802. PMID 7935655